CLINICAL TRIAL: NCT03902028
Title: Interest of an Optimized Medico-pharmaceutical Collaboration in the Drug Management of Patients With Heart Failure: Controlled, Randomized, Multicentric Study
Brief Title: Optimized Medico-pharmaceutical Collaboration in the Drug Management of Patients With Heart Failure
Acronym: COMPIC
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: RECHMPL18_0040
Record Dates: First submitted 2019-03-27; First posted 2019-04-03 (Actual); Last update posted 2022-01-04 (Actual); Status verified 2021-12

CONDITIONS: Heart Failure
Keywords: Heart failure; pharmacist; multidisciplinary team; readmission
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Reinforced multidisciplinary follow-up (Experimental): Entrance medication reconciliation performed by a pharmacist
  * Patient compliance evaluation
  * Patient quality of life evaluation
  * Pharmaceutical analysis with focus on medication optimization with a specific check-list (according to ESC 2016 recommendations)
  * Hospitalisation discharge medication reconciliation
  * Patient pharmaceutic interview at the hospitalisation discharge
  * Transmission of informations to the general practitioner and the pharmacist's patient
  * Multidisciplinary consult at 1 month after hospitalisation discharge
  Interventions: Other: Reinforced multidisciplinary follow-up
- Standard care (No Intervention): * Drug review by a paramedic or a pharmacist
  * Pharmaceutical analysis
  * Therapeutic optimisation based on the usual practices care of the cardiologic department
  * Writing of the prescription given on leaving hospital based on the usual care of the department
  * Treatments explanations and support to the patient on the usual care
  * Transmission of the hospitalisation report to the patient general practitioner as the usual practice
  * Medical consult in usual time frames (an average of 1 month after hospitalisation discharge) at the patient location of choice

INTERVENTIONS:
Other: Reinforced multidisciplinary follow-up — Reinforced multidisciplinary follow-up
  Arms: Reinforced multidisciplinary follow-up

SUMMARY:
This is a controlled, randomized, open-label, multicentric study evaluating the value of coordinated medico-pharmaceutical management compared to standard management in patients with heart failure. The aim of this study is to evaluate the impact of these optimized activities on the re-hospitalization of the patient with cardiac insufficiency for a disease-related event within three months of the initial hospitalization.

DETAILED DESCRIPTION:
Heart failure (FH) is a public health problem with an estimated prevalence of about 1.5% in developed countries. In 2013, the number of patients hospitalized in France for heart failure amounted to 165 231 and 20% of them were re-hospitalized at least once for the same reason during this year. Several factors contribute to the occurrence of cardiac decompensation (DC) : some modifiable (age, severity of IC, etiology ...) and others modifiable, such as therapeutics. Various elements could reduce the frequency of re-hospitalizations and the mortality due to this disease :

* a better knowledge of treatments by patients and consequently a better therapeutic compliance
* a better knowledge of the factors and signs of DC (low-sodium diet, weighing...)
* a better implementation of prescribing recommendations : less than 50% of patients have optimal treatment compared to ESC recommendations
* a better communication at the transition points of the patient pathway. The creation of a binomial cardiologist-clinical pharmacist during hospitalization and the maintenance of this optimized multidisciplinary follow-up within 3 months post-hospitalization is a proposal to intervene on these factors. Indeed, the clinical pharmacist (present in the care unit) works in collaboration with the medical and paramedical teams and can improve the care of patients. In the experimental group, a specific multidisciplinary consultation is planned for one month after the end of the hospitalization. A 3-month follow-up visit will be carried out by phone call to meet the criteria for readmission, mortality, quality of life, adherence and persistence of treatments.

ELIGIBILITY:
Inclusion Criteria:

* Patient aged more than 18 years
* Adult patient admitted in cardiology department (full hospitalisation or intensive care) for heart failure no matter the type and the stage of the disease
* Person affiliated or beneficiary of a social security system
* Collection of a free, informed, express and written consent

Exclusion Criteria:

* Non autonomous drug management patients and not disposing
* a present caregiver during hospitalisation
* Patients living in an institution
* Person participating in another clinical trial with an exclusion period still ongoing
* Person whose physical and/or psychological health is severely altered, and which, in the opinion of the investigator, may affect the participation's to the study
* Person deprived of his rights, person under tutorship or guardianship
* Refusal to sign the consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 248 (Estimated)
Dates: Start 2019-08-02 (Actual); Primary Completion 2022-02 (Estimated); Study Completion 2022-08 (Estimated)

PRIMARY OUTCOMES:
Rehospitalisation for heart failure | Call at 3 months after hospitalisation discharge
  At least one rehospitalisation with heart failure related cause

SECONDARY OUTCOMES:
Prescriptions conformity rates compared to heart failure recommendations edited by the European Society of Cardiology in 2016 | At hospitalisation discharge (Day 0)
  Evaluated by a pharmacist
Prescriptions conformity rates compared to heart failure recommendations edited by the European Society of Cardiology in 2016 | Call at 3 months after hospitalisation discharge
  Evaluated by a pharmacist
Compliance level | At hospitalisation discharge (Day 0)
  Evaluated by the " Girerd medication adherence questionnaire "
  The " Girerd medication adherence questionnaire " contains 6 questions which answers are " yes " or " no ". The number of " yes " responses permits to evaluate the level of the patient medication adherence as following :
  0 yes : good compliance
  1 or 2 yes : minor non compliance 3 or more yes : non compliance
Compliance level | At 1 month after hospitalisation discharge for the experimental group only
  Evaluated by the "Girerd medication adherence questionnaire" Evaluated by the " Girerd medication adherence questionnaire "
  The " Girerd medication adherence questionnaire " contains 6 questions which answers are " yes " or " no ". The number of " yes " responses permits to evaluate the level of the patient medication adherence as following :
  0 yes : good compliance
  1 or 2 yes : minor non compliance 3 or more yes : non compliance
Compliance level | Call at 3 months after hospitalisation discharge
  Evaluated by the "Girerd medication adherence questionnaire" Evaluated by the " Girerd medication adherence questionnaire "
  The " Girerd medication adherence questionnaire " contains 6 questions which answers are " yes " or " no ". The number of " yes " responses permits to evaluate the level of the patient medication adherence as following :
  0 yes : good compliance
  1 or 2 yes : minor non compliance 3 or more yes : non compliance
Treatment persistence rates | Call at 3 months after hospitalisation discharge
  Evaluated by a pharmacist
Death rate | Call at 3 months after hospitalisation discharge
  Evaluated by a pharmacist
Time before death | Call at 3 months after hospitalisation discharge
  Evaluated by a pharmacist
Time of occurrence of a potential rehospitalisation related to the disease | Call at 3 months after hospitalisation discharge
  Evaluated by a pharmacist
Quality of life score | Call at 3 months after hospitalisation discharge
  Evaluated by the Minnesota Living with Heart Failure Questionnaire the Minnesota Living with Heart Failure Questionnaire contains 21 questions. Each of the 21 questions ask the patients to indicate how much a possible effect of heart failure have affected their ability to live as wanted during the past month using a scale from 0 (not present or no effect), 1 (very little), 2, 3, 4, or 5 (very much).The measurement of heart failure severity is assessed by summing the responses that ranges from 0 to 105.
Satisfaction of the patient | Call at 3 months after hospitalisation discharge
  Evaluated by Likert scale This questionnaire indicates the degree of patient satisfaction using 9 questions which explore the improvement of patient behavior concerning disease and treatment. The measurement of satisfaction is assessed by summing the responses that range from 9 (unsatisfied) to 36 (very satisfied)
Satisfaction of health professionals | online questionnaire at 3 months after hospitalisation discharge
  Evaluated by Likert scale (only for interventional arm) This questionnaire indicates the degree of health professional satisfaction using 6 questions which explore the improvement of transition between hospital to community and comprehension of therapeutic optimization. The measurement of satisfaction is assessed by summing the responses that range from 6 (unsatisfied) to 24 (very satisfied)
Incremental cost-effectiveness ratio | 3 months after hospitalisation discharge

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital of Montpellier Cardiology departments oh the Montpellier, Nîmes and Toulouse University Hospitals, Montpellier, Occitanie, France

REFERENCES:
- [Result] Jackevicius CA, de Leon NK, Lu L, Chang DS, Warner AL, Mody FV. Impact of a Multidisciplinary Heart Failure Post-hospitalization Program on Heart Failure Readmission Rates. Ann Pharmacother. 2015 Nov;49(11):1189-96. doi: 10.1177/1060028015599637. Epub 2015 Aug 10. PMID 26259774
- [Result] Ponikowski P, Voors AA, Anker SD, Bueno H, Cleland JGF, Coats AJS, Falk V, Gonzalez-Juanatey JR, Harjola VP, Jankowska EA, Jessup M, Linde C, Nihoyannopoulos P, Parissis JT, Pieske B, Riley JP, Rosano GMC, Ruilope LM, Ruschitzka F, Rutten FH, van der Meer P; ESC Scientific Document Group. 2016 ESC Guidelines for the diagnosis and treatment of acute and chronic heart failure: The Task Force for the diagnosis and treatment of acute and chronic heart failure of the European Society of Cardiology (ESC)Developed with the special contribution of the Heart Failure Association (HFA) of the ESC. Eur Heart J. 2016 Jul 14;37(27):2129-2200. doi: 10.1093/eurheartj/ehw128. Epub 2016 May 20. No abstract available. PMID 27206819
- [Result] Available at: https://academic.oup.com/eurheartj/article/37/27/2129/1748921/2016-ESC-Guidelines-for-the-diagnosis-and. (Accessed: 12th September 2017).
- [Result] Masters J, Morton G, Anton I, Szymanski J, Greenwood E, Grogono J, Flett AS, Cleland JG, Cowburn PJ. Specialist intervention is associated with improved patient outcomes in patients with decompensated heart failure: evaluation of the impact of a multidisciplinary inpatient heart failure team. Open Heart. 2017 Mar 8;4(1):e000547. doi: 10.1136/openhrt-2016-000547. eCollection 2017. PMID 28409010
- [Result] Van Spall HGC, Rahman T, Mytton O, Ramasundarahettige C, Ibrahim Q, Kabali C, Coppens M, Brian Haynes R, Connolly S. Comparative effectiveness of transitional care services in patients discharged from the hospital with heart failure: a systematic review and network meta-analysis. Eur J Heart Fail. 2017 Nov;19(11):1427-1443. doi: 10.1002/ejhf.765. Epub 2017 Feb 24. PMID 28233442
- [Result] Lopez Cabezas C, Falces Salvador C, Cubi Quadrada D, Arnau Bartes A, Ylla Bore M, Muro Perea N, Homs Peipoch E. Randomized clinical trial of a postdischarge pharmaceutical care program vs regular follow-up in patients with heart failure. Farm Hosp. 2006 Nov-Dec;30(6):328-42. doi: 10.1016/s1130-6343(06)74004-1. English, Spanish. PMID 17298190
- [Result] Parajuli DR, Franzon J, McKinnon RA, Shakib S, Clark RA. Role of the Pharmacist for Improving Self-care and Outcomes in Heart Failure. Curr Heart Fail Rep. 2017 Apr;14(2):78-86. doi: 10.1007/s11897-017-0323-2. PMID 28233258
- [Result] Wan TTH, Terry A, Cobb E, McKee B, Tregerman R, Barbaro SDS. Strategies to Modify the Risk of Heart Failure Readmission: A Systematic Review and Meta-Analysis. Health Serv Res Manag Epidemiol. 2017 Apr 18;4:2333392817701050. doi: 10.1177/2333392817701050. eCollection 2017 Jan-Dec. PMID 28462286
- [Result] Buckley MS, Harinstein LM, Clark KB, Smithburger PL, Eckhardt DJ, Alexander E, Devabhakthuni S, Westley CA, David B, Kane-Gill SL. Impact of a clinical pharmacy admission medication reconciliation program on medication errors in "high-risk" patients. Ann Pharmacother. 2013 Dec;47(12):1599-610. doi: 10.1177/1060028013507428. Epub 2013 Oct 15. PMID 24259613
- [Result] Warden BA, Freels JP, Furuno JP, Mackay J. Pharmacy-managed program for providing education and discharge instructions for patients with heart failure. Am J Health Syst Pharm. 2014 Jan 15;71(2):134-9. doi: 10.2146/ajhp130103. PMID 24375606